CLINICAL TRIAL: NCT07045753
Title: A Prospective Follow-up Assessment in Bad Segeberg With Patients With Severe Mitral Regurgitation Undergoing Mitral Edge-to-edge Repair (M-TEER).
Brief Title: The Prospective Segeberg Registry for Mitral Transcatheter Edge-to-Edge Repair
Acronym: SK M-CLIP
Status: Recruiting | Type: Observational
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SK 113 - 168/11
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Mitral Regurgitation (MR)
Keywords: M TEER; Mitral Clip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of severe MR undergoing M-TEER: Patients with severe mitral regurgitation undergoing transcatheter edge to edge repair (M-TEER)
  Interventions: Device: Transcatheter edge to edge repair

INTERVENTIONS:
Device: Transcatheter edge to edge repair — mitral valve transcatheter edge-to-edge repair
  Other Names: M TEER; Mitral Clip

SUMMARY:
A Prospective Follow-up Assessment in Bad Segeberg for Patients with severe MR undergoing M-TEER

DETAILED DESCRIPTION:
A prospective single center registry including all patients treated for severe mitral regurgitation (MR) with mitral edge-to-edge repair (M-TEER) at the Heart Center, Bad Segeberg, Germany. Patients undergo a routine clinical follow-up schedule, including a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe MR undergoing M-TEER

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe MR undergoing M-TEER
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of in-hospital and long-term cardiovascular adverse events in percent | 2 years
  Peri-procedural events and in-hospital cardiovascular events and long-term cardiovascular events (bleeding, peripheral and coronary vascular complication, stroke, myocardial infarction, stent thrombosis, revascularization, death, heart failure, rehospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Nef, Prof., MD, Study Director — Herzzentrum Segeberger Kliniken GmbH
Locations (1):
- Herzzentrum Segeberger Kliniken GmbH, Bad Segeberg, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No